CLINICAL TRIAL: NCT06399055
Title: A Randomized, Open-label, Single Dose, Crossover Study to Evaluate the Pharmacokinetic Profiles and Safety of CKD-387 in Healthy Volunteers Under Fasting Conditions
Brief Title: Clinical Study to Evaluate the Pharmacokinetic Profiles and Safety of CKD-387 in Healthy Volunteers Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A84_08BE2207
Record Dates: First submitted 2024-01-22; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Endocrine, Nutritional and Metabolic Diseases
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference-Test (Experimental)
  Interventions: Drug: CKD-387; Drug: D484
- Test- Reference (Experimental)
  Interventions: Drug: CKD-387; Drug: D484

INTERVENTIONS:
Drug: CKD-387 — 1 Tablet
  Other Names: Test
Drug: D484 — 1 Tablet
  Other Names: Reference

SUMMARY:
This study is a randomized, open-label, single dose, crossover study to evaluate the pharmacokinetic profiles and safety of CKD-387 in healthy volunteers under fasting conditions.

DETAILED DESCRIPTION:
To 36 healthy subjects, following treatments are administered dosing in each period and wash-out period is a minimum of 7 days Pharmacokinetic blood samples are collected up to 48hrs. The pharmacokinetic characteristics and safety are assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults volunteers aged between 19 and 55 years old at the time of screening
2. Individuals who had 17.5 kg/m2 ≤ Body Mass Index(BMI) < 30.5kg/m2 and men's total body weight ≥ 55 kg, women's total body weight ≥ 45 kg

   * BMI = Weight(kg)/ Height(m)2
3. Individuals without congenital/chronic diseases and without abnormal symptoms or diagnosis based on a medical examination within the last 3 years
4. Individuals who were deemed to be appropriate as study subjects following laboratory tests (hematology, blood chemistry, urinalysis, viral/bacterial, etc.) and vital signs, ECG etc. performed at screening
5. Individuals who signed an informed consent form approved by the Institutional Review Board of Bumin Hospital and decided to participate in the study after being fully informed of the study prior to participation, including the objective and content
6. Individuals who agreed proper contraception during the study and did consent to not donation of sperm 1 month after the last dose of study drug infusion
7. Individuals with the ability and willingness to participate the entire study period

Exclusion Criteria:

1. Individuals with a medical evidence or a history (excluding a dental history of periodontal surgery, impacted wisdom teeth removal, etc.) of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, urinary, cardiovascular, hepatic, psychiatric, neurologic or immune diseases.
2. Individuals with a medical history of gastrointestinal disease (e.g., gullet disease such as esophageal achalasia and esophagostenosis and Crohn's disease) or operations (excluding simple appendectomy, herniotomy or tooth extraction) that may affect drug absorption
3. Individuals with the following laboratory test results at screening:

   - Alanine aminotransferase or Aspartate transaminase > 2x the upper limit of the normal range
4. History of regular alcohol consumption exceeding 210 g/week within the 6 months prior to screening (1 drink (250 mL) of beer (5%) = 10 g; 1 drink (50 mL) of hard liquor (20%) = 8 g; 1 drink (125 mL) of wine (12%) = 12 g)
5. Individuals who smoked more than 20 cigarettes per day within 6 months or consumed more than 5 cups of caffeine per day prior to first administration of investigational drugs
6. Individuals who had been administered investigational product(s) from other clinical study or bioequivalence study within the 6 months prior to the first administration of investigational drugs
7. Following vital signs results at screening

   - Sitting systolic blood pressure ≥ 150 mmHg or < 90 mmHg and/or sitting diastolic blood pressure ≥100 mmHg or <50 mmHg
8. Individuals with a medical history of significant alcohol or drug abuse within one year prior to the screening
9. Individuals who had taken any drug(s) known as a strong inducer(s) or inhibitor(s) of drug-metabolizing enzymes within 30 days prior to the first administration of investigational drugs
10. Individuals who had taken prescription or nonprescription drugs within the 10 days prior to the first administration of investigational drugs
11. Individuals who donated whole blood within the 8 weeks, or blood components within 2 weeks prior to the first administration of investigational drugs
12. Individuals with severe acute/chronic medical or psychiatric condition that may increase the risk associated with study participation or investigational product(s) administration, or may interfere with the interpretation of study results
13. Individuals with hypersensitivity to investigational products or the investigational products ingredients
14. Patients with nephropathy (eGFR<60 ml/min/1.73 m2)
15. Acute conditions that can affect renal function such as dehydration, severe infection, cardiovascular collapse (shock), acute myocardial infarction, and sepsis
16. Patients with acute or chronic metabolic acidosis including type 1 diabetes mellitus, lactic acidosis, or diabetic ketoacidosis with or without coma, and patients with a history of ketoacidosis
17. Diabetic precoma
18. Patients undergoing intravenous administration of radioactive iodine contrast material (e.g., intravenous urography, venous cholangiography, angiography, computed tomography using contrast medium, etc.)
19. Patients with congestive heart failure or heart failure who require drug treatment (NYHA class IV)
20. Patients with severe infection or severe traumatic systemic disorder
21. Patients with malnutrition, starvation, weakness, pituitary insufficiency or adrenal insufficiency
22. Patients with genetic problems such as galactose intolerance, Lap lactase deficiency, or glucose-galactose malabsorption
23. Women who are pregnant or may be pregnant
24. Individuals who were deemed to be inappropriate to participate in the study by the investigator

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-10-09 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-387, D484 | (Pre-dose) 0 hour, (Post-dose) 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48 hours
  Area under the CKD-387, D484 concentration in blood-time curve from 0 to last sampling time (t)
Cmax of CKD-387, D484 | (Pre-dose) 0 hour, (Post-dose) 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48 hours
  The maximum CKD-387, D484 concentration in blood sampling time (t)

CONTACTS AND LOCATIONS:
Locations (1):
- Bumin Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No